The Effect of Immediate Versus Delayed Debriefing on Basic Life Support Competence In Undergraduate Nursing Students.

NCT06624449 October 5, 2023

Alanezi, Fahad (alanezfz)

[Company Name] | [Company Address]

The statistical analysis was conducted using JMP Pro 16 software. Descriptive statistics for the students' demographics were calculated, including means, standard deviations, and frequencies. A Paired t-test was used to determine the differences between the experimental and control groups before and after the intervention. An independent t-test was applied to examine differences in BLS competence levels between the two groups. A p-value of less than 0.05 was considered statistically significant, with a 95% confidence interval. If the p-value was below 0.05, the null hypothesis would be rejected; if it exceeded 0.05, we would fail to reject the null hypothesis. Independent t-tests were also used to compare the mean debriefing experience scores between the hot and cold debriefing groups, with p-values below 0.05 considered statistically significant.